CLINICAL TRIAL: NCT02367677
Title: Comparison Between Clinical Measurements and Computer-based Measurements on Digital Photographs to Evaluate Blepharoptosis
Brief Title: Digital Photographs to Evaluate Blepharoptosis
Status: Completed | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-1905, C14-06-1905
Record Dates: First submitted 2015-02-03; First posted 2015-02-20 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-08

CONDITIONS: Blepharoptosis
Keywords: Photo
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Clinical measurements: Measurements are made with a paper ruler
  Interventions: Other: Method comparison
- Smartphone: Measurements are made with ImageJ from pictures taken with an iPhone 6
  Interventions: Other: Method comparison
- Digital camera: Measurements are made with ImageJ from pictures taken with a Nikon D700
  Interventions: Other: Method comparison

INTERVENTIONS:
Other: Method comparison

SUMMARY:
To compare measurements made by a computer software (ImageJ) made on photographs to the traditional clinical measures with a ruler in the evaluation of blepharoptosis

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older
* Patients presenting for evaluation of blepharoptosis of any kind except the one mentioned in the exclusion criteria

Exclusion Criteria:

* Myasthenia gravis
* Thyroid eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ptosis of all causes
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Reliability of measurements made on photographs to evaluate blepharoptosis | Same day
  Comparison between measurements made on digital photographs with measurements made with a ruler in clinic
Reliability of measurements made on photographs taken by smartphone to evaluate blepharoptosis | Same day
  Comparison between measurements made on digital photographs taken by smartphone with measurements made on digital photographs taken with a digital camera

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Molgat, MDCM, FRCSC, Principal Investigator — Centre de recherche du CHU de Québec : Université Laval
Locations (1):
- Centre Universitaire d'Ophtalmologie, Hôpital du Saint-Sacrement, CHU de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided